CLINICAL TRIAL: NCT05416697
Title: Effectiveness of Cannabinoid on Appetite, Sleep Quality, Quality of Life, Joint Pain, and Cytokine Level in Systemic Sclerosis Patients: a Randomized Placebo-controlled Trial
Brief Title: Effectiveness of Cannabinoids on Appetite in Scleroderma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Chingching Foocharoen, Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cannabinoid in scleroderma
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Systemic Sclerosis; Malnutrition; Loss of Appetite
Keywords: cannabinoid; appetite; quality of life; systemic sclerosis; scleroderma; clinical trial
MeSH Terms: conditions — Scleroderma, Systemic; Malnutrition; Anorexia; Scleroderma, Diffuse

STUDY DESIGN:
Intervention Model Description: cannabinoid versus placebo
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participant, care provider, and assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cannabinoid (Experimental): Cannabinoid in form of cannabis 2.7 mg THC 2.5 mg twice daily (1 droplet twice daily; 0.73 mg THC and 0.81 mg CBD/drop, 1.46 mg THC and 1.62 CBD/day) for 1 week then titrate up to 2 droplets twice daily if tolerated (2.92 mg THC and 3.24 CBD per day) and continue the treatment until the end of the study
  Interventions: Drug: CBD oil
- placeba (Placebo Comparator): Placebo 1 droplet twice daily for 1 week then titrate up to 2 droplets twice daily if tolerated and continue the treatment until the end of the study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBD oil — The subjects will receive cannabis 2.7 mg THC 2.5 mg CBD twice daily (1 droplet twice daily; 0.73 mg THC and 0.81 mg CBD/drop, 1.46 mg THC and 1.62 CBD/day) for 1 week then titrate up to 2 droplets twice daily if tolerated (2.92 mg THC and 3.24 CBD per day) and continue the treatment until the end of the study.
  Arms: cannabinoid
Drug: Placebo — The subjects will receive 1 droplet of placebo twice daily then titrate up to 2 droplets twice daily if tolerated and continue the treatment until the end of the study.
  Arms: placeba

SUMMARY:
The cannabinoid has benefits in many aspects but the evidence of the effect of cannabinoids in humans with SSc is limited. We, therefore, would like to investigate the efficacy of cannabinoids on the appetite, sleep efficiency, quality of life, pain, and critical cytokine level in SSc compared with placebo in SSc patients and the adverse events associated with cannabinoids in those patients.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a connective tissue disease for which skin tightness is the hallmark. The disease is classified into 2 major subsets: limited cutaneous systemic sclerosis (lcSSc) and diffuse cutaneous systemic sclerosis (dcSSc) depending on the extent of skin tightness. Not only the skin tightness but also the internal organs such as the musculoskeletal, kidneys, lungs, heart, and intestines can be involved and associated with a poor outcome. Malnutrition and/or weight loss is a complications in SSc. The complication is possibly related to gastrointestinal involvement, inflammation, immunosuppressant agents, or mood disturbance which can affect the food appetite or eating behavior. As well as sleep quality, sleep disturbance has been reported in SSc patients and the associated factor of sleep disturbance in those patients was gastrointestinal involvement, particularly gastroesophageal reflux disease, the severity of pain, and depressed mood. The cannabinoid is an agent which affects appetite, pain, and sleep quality as mentioned above, hence it would improve the appetite, get a high sleep quality and reduce pain associated with musculoskeletal involvement in SSc patients.

Although cannabinoid has benefit in many aspects, they also resulted in serious adverse events after cannabinoid inhalation, including ischemic stroke related to vasospasm of the cerebral vessel, high cardiac output, cardiac arrhythmias, blood pressure fluctuation, and respiratory tract infection. Acute toxicity has been reported and depended on unit dose, tolerance, and route of cannabinoid use. Cannabis also influenced brain function including memory, and cognitive function, and expanded the risk for psychosis in those who had prolonged use. The symptoms of central nervous system (CNS) toxicity include euphoria, panic, agitation, mood alterations, alteration of perception, loss of social inhibition, muscle incoordination, myoclonic jerking, ataxia, slurred speech, and risk of the suicidal idea. In addition, prolonged high doses of cannabis use can lead to the development of cannabinoid hyperemesis syndrome caused by cyclic hyperemesis, finally resulting in electrolyte disturbances and impaired kidney function.

Because the evidence of the effect of cannabinoids in humans with SSc is limited. We, therefore, would like to investigate the efficacy of cannabinoids on the appetite, sleep efficiency, quality of life, pain, and key cytokine level in SSc compared with placebo in SScpatientst and the adverse events associated with cannabinoids in those patients.

ELIGIBILITY:
Inclusion Criteria:

1. SSc patients aged between 18 and 70 years
2. Diagnosed according to ACR/EULAR 2013 classification criteria
3. Having anorexia or malnutrition status
4. Must not receive steroid equivalent to prednisolone dose more than 10 mg/d
5. Must receive a stable dose of steroid, immunosuppressant, and/or vitamin or its supplement within 2 weeks before enrollment
6. Must stop anxiolytics, hypnotics, or sleeping pills at least 2 weeks before enrollment
7. Understand and able to read and write the Thai language

Exclusion Criteria:

1. Overlap with other connective tissue diseases
2. Pregnancy or lactation
3. Bedridden and confined to no self-care
4. Evidence of active malignant disease
5. Present uncontrolled or severe medical problems including diabetes mellitus, asthma, angina, cardiovascular, thyroid, hepatic, or renal diseases (Cr>1.4 mg/dl)
6. Present active infection that needs systemic antibiotic
7. Previous allergy to cannabinoid or their derivatives
8. Concomitant illegal drug used (amphetamine or its derivative, cocaine)
9. History of the previous cannabinoid using or concomitant any herbal included cannabinoid used
10. On-going anxiolytics, hypnotics, or sleeping pills used
11. In a period that needs immunosuppressant dose adjustment
12. Having active SSc that needs closed monitoring for disease progression (pulmonary hypertension, proteinuria, microscopic hematuria, digital gangrene, and progressive interstitial lung disease)
13. Having unstable cardiopulmonary disease (angina, peripheral vascular disease, cerebrovascular disease, and arrhythmia) and risk of cardiovascular disease
14. Having a history of schizophrenia, concurrent active mood disorder, or anxiety disorders
15. Receiving the following medications that cause drug interaction with cannabinoids: fluoroquinolone, rifampicin, fluoxetine, warfarin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The changing of appetite | 4 weeks
  50% increase of appetite evaluated by a visual analogue scale (VAS) from 0-100* compared to baseline and a comparison between the treatment group and placebo group
  *a higher score, a more appetite

SECONDARY OUTCOMES:
The changing of serum transferrin level | 4 weeks
  The mean difference of serum transferrin level compare to baseline and a comparison between the treatment group and placebo group
An adverse event | 4 weeks
  An adverse event

OTHER OUTCOMES:
The changing of sleep quality | 4 weeks
  The changing of sleep quality evaluated by the Thai Pittsburgh Sleep Quality Index* compare to baseline and a comparison between the treatment group and placebo group
  *the score ranges from 0-to 21 and the higher score, the poorer sleep quality
The changing of quality of life | 4 weeks
  The changing of the quality of life evaluated by EuroQol group 5 dimensions (EQ-5D)* compare to baseline and a comparison between the treatment group and placebo group
  *the index composes of 5 dimensions and each dimension includes 3 levels (no problems, some problems, and extreme problems), the higher level of the dimension, the poorer quality of life
The changing pain symptoms | 4 weeks
  50% decrease of joint pain evaluated by VAS from 0-100* compare to baseline and a comparison between the treatment group and placebo group
  *a higher scale, a more pain
The changing of cytokine level (transforming growth factor beta) | 4 weeks
  The changing of cytokine level compare to baseline and a comparison between the treatment group and placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Chingching Foocharoen, M.D., Principal Investigator — Khon Kaen University
Locations (2):
- Thailand (2):
  - Department of Medicine, Faculty of Medicine, Khon Kaen University, Khon Kaen
  - Scleroderma Clinic, Faculty of Medicine, Khon Kaen University, Khon Kaen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pisprasert V, Sripanichkulchai B, Khannongpho T, Jumnainsong A, Mahakkanukrauh A, Suwannaroj S, Pongkulkiat P, Onchan T, Kanokmedhakul S, So-Ngern A, Foocharoen C. Efficacy of cannabis oil on appetite and quality of life in systemic sclerosis patients: a randomized placebo-controlled trial. J Cannabis Res. 2025 Oct 24;7(1):82. doi: 10.1186/s42238-025-00342-3. PMID 41137182